CLINICAL TRIAL: NCT04794270
Title: Evaluation of ACUVUE OASYS® 1-Day for Astigmatism Lenses Produced on a New Manufacturing Line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6420
Record Dates: First submitted 2021-02-19; First posted 2021-03-12 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized into the (TEST/CONTROL) sequence and will wear two different study lenses one at a time over the two wear periods. During each wear period the lenses will be worn bilaterally for approximately 1 week. Study lenses will be worn for a minimum of 8 hours per day and at least 5 days per week during the wear period.
  Interventions: Device: ACUVUE OASYS® 1-Day for Astigmatism - TAM 24; Device: ACUVUE OASYS® 1-Day for Astigmatism
- CONTROL/TEST (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized into the (CONTROL/TEST) sequence and will wear two different study lenses one at a time over the two wear periods. During each wear period the lenses will be worn bilaterally for approximately 1 week. Study lenses will be worn for a minimum of 8 hours per day and at least 5 days per week during the wear period.
  Interventions: Device: ACUVUE OASYS® 1-Day for Astigmatism - TAM 24; Device: ACUVUE OASYS® 1-Day for Astigmatism

INTERVENTIONS:
Device: ACUVUE OASYS® 1-Day for Astigmatism - TAM 24 — TEST
Device: ACUVUE OASYS® 1-Day for Astigmatism — CONTROL

SUMMARY:
This is a bilateral, dispensing, randomized, controlled, double-masked, 2×2 cross-over study to evaluate the clinical performance of ACUVUE OASYS® 1-Day for Astigmatism contact lenses produced on a recently qualified manufacturing line.

ELIGIBILITY:
Inclusion Criteria:

- Potential subjects must satisfy all of the following criteria to be enrolled in the study:

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 2 days per week during the past month.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. Have the spherical component of their vertex-corrected distance refraction must be between -0.875 to -4.625 DS (inclusive) in each eye.
7. Have the magnitude of the cylindrical component of their vertex-corrected distance refraction between 0.625 DC and 1.625 DC in both eyes.
8. Have the cylinder axis of their distance refraction between 165° and 15° (i.e., 180±15°, inclusive) or between 75° and 105° (i.e., 90±15°, inclusive) in each eye.
9. Have best corrected monocular distance visual acuity of 20/30 or better in each eye.

Exclusion Criteria:

- Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have any ocular infection of any type.
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses.
7. Be currently wearing lenses in an extended wear modality.
8. Have a history of strabismus or amblyopia.
9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (5):
- United States (5):
  - Sabal Eye Care, Longwood, Florida
  - VisionPoint Eye Center, Bloomington, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - Sacco Eye Group, Vestal, New York
  - Professional Vision Care, Inc., Westerville, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 72 subjects were enrolled in this study. Of those enrolled, a total of 71 subjects were assigned to one of two wear sequences; while one subject was a screen failure and/or not assigned. Of the total assigned subjects, 68 subjects completed the study while, 3 subjects were discontinued from the study.
Groups:
- Control/Test: Subjects that wore the Control lens in a bilateral fashion during Period 1 and the Test lens during Period 2.
- Test/Control: Subjects that wore the Test lens in a bilateral fashion during Period 1 and the Control lens during Period 2.
Period: Period 1
Arm/Group | Control/Test | Test/Control
Started | 35 | 36
Completed | 33 | 36
Not Completed | 2 | 0
Not completed — Non Compliance | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2
Arm/Group | Control/Test | Test/Control
Started | 33 | 36
Completed | 32 | 36
Not Completed | 1 | 0
Not completed — Unsatisfactory Lens Fitting due to Test Article | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study article.
Groups:
- Dispensed Subject: All subjects dispensed a study article.
Arm/Group | Dispensed Subject
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Black or African American | 2
  White | 67
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: CLUE Comfort Score
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: Fitting, 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Test: All subjects that wore the Test lens during any of the 2 wear periods.
- Control: All subjects that wore the Control lens during any of the 2 wear periods.
Arm/Group | Test | Control
Number analyzed (Participants) | 58 | 58
Units on a scale
  Fitting | 65.95 (18.645) | 65.13 (18.849)
  1-Week Follow-up | 67.39 (20.024) | 70.80 (22.742)

2. Primary Outcome: CLUE Vision Score
Description: Overall vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: Fitting, 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test | Control
Number analyzed (Participants) | 58 | 58
Units on a scale
  Fitting | 70.14 (15.979) | 69.64 (15.767)
  1-Week Follow-up | 68.33 (18.349) | 72.40 (19.381)

3. Primary Outcome: CLUE Handling Score
Description: Overall handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: Fitting, 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test | Control
Number analyzed (Participants) | 58 | 58
Units on a scale
  Fitting | 73.56 (19.057) | 72.71 (20.760)
  1--Week Follow-up | 70.61 (21.048) | 71.83 (19.740)

4. Primary Outcome: Monocular Visual Performance (LogMAR)
Description: Visual performance was calculated as monocular contact lens-corrected distance visual acuity using a Logarithm of Minimal Angle of Resolution (logMAR) visual acuity scale. This was evaluated under high luminance and high contrast conditions (HLHC) at 4 meters from Early Treatment Diabetic Retinopathy Study (ETDRS) charts at the 1-week follow-up visit. Lower visual performance values indicate better vision. Two measurements were performed for each eye. The average visual performance was reported for each lens type.
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eye
Arm/Group | Test | Control
Number analyzed (Participants) | 58 | 58
Number analyzed (eye) | 116 | 116
LogMAR | -0.108 (0.0703) | -0.112 (0.0679)

5. Primary Outcome: Lens Rotation
Description: Lens rotation was recorded from direction and magnitude in degrees to the nearest degree at one and three minutes following lens insertion during settling period. All lenses in this study have scribe marks at 6 o'clock and 12 o'clock positions and rotation measurements were made relative to a vertical reference line.
Time Frame: Post-Fitting at 1-minute, at 3-minute
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: eye
Arm/Group | Test | Control
Number analyzed (Participants) | 58 | 58
Number analyzed (eye) | 116 | 116
Degrees
  At 1-minute | -1.7 (14.65) | -2.0 (14.94)
  At 3-minute | -1.1 (4.55) | -0.8 (4.88)

6. Primary Outcome: Settled Rotation
Description: Mean settled rotation was calculated from all repeated measures of signed lens orientation upon settling for each subject/eye/lens.
Time Frame: Fitting, 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: eye
Arm/Group | Test | Control
Number analyzed (Participants) | 58 | 58
Number analyzed (eye) | 116 | 116
Degrees
  Fitting | -0.9 (2.69) | -1.3 (2.80)
  1-Week Follow-up | -1.8 (3.29) | -1.6 (3.26)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 3 weeks per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 0/71 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT04794270/Prot_SAP_000.pdf